CLINICAL TRIAL: NCT01712035
Title: OCT Evaluation of Treated and Untreated Choroidal Neovascular Membranes in Age-Related Macular Degeneration
Brief Title: Neovascular Age-related Macular Degeneration
Acronym: NVAMD
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Steven T. Bailey, MD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: OHSU IRB #00008360
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Wet AMD; Age-related macular degeneration; Optical coherenece tomography; Imaging; Blood flow
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Treatment-active NVAMD: Patients with NVAMD who have received treatment with an anti-VEGF agent (Avastin, Lucentis, Macugen, or Eylea) 6 weeks prior enrollment visit
- Treatment-naive NVAMD: Individuals who have not received any treatment for neovascular AMD in the study eye

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of blindness in non-Hispanic white Americans. Neovascular AMD is an advanced form of macular degeneration that historically has accounted for the majority of vision loss related to AMD. The presence of choroidal neovascular membrane (CNV) formation is the hallmark feature of neovascular AMD. Choroidal neovascular membranes consist of buds of neovascular tissue and accompanying fibroblasts from the choroid perforating Bruch's membrane with extension either above or below the retinal pigment epithelium. These neovascular complexes are associated with hemorrhage, fluid exudation and fibrosis formation resulting in photoreceptor damage and vision loss. Treatment of neovascular AMD consists of injecting inhibitors of vascular endothelial growth factor (VEGF) into the vitreous cavity to interfere with proliferation of choroidal neovascularization and to reduce vascular permeability.

OCT is an imaging technology that can perform non-contact cross-sectional imaging of retinal and choroidal tissue structure in real time. It is analogous to ultrasound B-mode imaging, except that OCT measures the intensity of reflected light rather than acoustical waves.

This observational study will use OCT technology to study and compare the retinal and choroidal anatomy and blood flow in two groups of patients with neovascular AMD: treatment naïve group and active treatment group.

The purpose of this study is to assess the utility of OCT angiography in the evaluation of NVAMD.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Neovascular AMD confirmed by fluorescein dye leakage on angiogram or presence of at least one of the following on OCT: subretinal fluid, intraretinal fluid, or sub-retinal pigment epithelial fluid.
* Treatment naïve group consists of individuals who have not received any treatment for neovascular AMD in the study eye
* Active treatment group consists of individuals who have received treatment with an anti-VEGF agent (Avastin, Lucentis, Macugen, or Eylea) 6 weeks prior enrollment visit

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
* Women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months due to unknown safety of fluorescein angiography.
* Unable to ambulate and take tram from clinic to where OCT is located
* Prior macular laser treatment
* Subretinal hemorrhage or fibrosis >50% of choroidal neovascular lesion
* Visual acuity 20/200 or worse
* An ocular condition is present such that, in the opinion of the investigator, may alter the retinal anatomy (eg: epiretinal membrane)
* An ocular condition is present (other than Neovascular AMD) that, in the opinion of the investigator, might affect or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, etc.).
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults older than age 50 with clinical findings of neovascular AMD with clinical evidence of active choroidal neovascular membrane
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with NVAMD receiving treatment who also have changed retinal/choroidal anatomy and/or blood flow compared to treatment naive NVAMD patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States